CLINICAL TRIAL: NCT02979210
Title: Fecal Insult Study: An Exploratory Study to Evaluate the Microbial Consortia and Skin Barrier Function After Exposure to Artificial Fecal Irritants
Brief Title: Infant Fecal Insult Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 500-16-0003
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial Fecal Insult (Other): protease/bile acid cocktail 200 microliters (1500 µg/ml trypsin/chymotrypsin protease mixture, 6.5 mg/ml cholic acid sodium, 6.2 mg/ml deoxycholic acid sodium, and 3.1 mg/ml chenodeoxycholic acid sodium in phosphate buffered saline)
  Interventions: Other: Artificial Fecal Insult; Other: Phosphate Buffered Saline

INTERVENTIONS:
Other: Artificial Fecal Insult — protease/bile acid cocktail 200 microliters (1500 µg/ml trypsin/chymotrypsin protease mixture, 6.5 mg/ml cholic acid sodium, 6.2 mg/ml deoxycholic acid sodium, and 3.1 mg/ml chenodeoxycholic acid sodium in phosphate buffered saline
Other: Phosphate Buffered Saline — 200 microliters of phosphate buffered saline

SUMMARY:
The rationale for the study is to better understand the dynamics of skin microflora following skin barrier disruption in an adult dermatitis model. The results from this study will provide insights in the complex interaction between skin microbiome and epidermis under normal and disease conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects with Fitzpatrick Skin Types I, II or III

Exclusion Criteria:

* Subjects with visible skin disease, tattoos, skin condition, or abnormal skin color

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01-26 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Type of microbes present on skin after exposure to artificial fecal insult | up to 7 days
  Microbes will be identified by metagenomic sequencing
Relative abundance of microbes present on skin measured in picograms of DNA | up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Reliance Clinical Testing Service, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Costello EK, Lauber CL, Hamady M, Fierer N, Gordon JI, Knight R. Bacterial community variation in human body habitats across space and time. Science. 2009 Dec 18;326(5960):1694-7. doi: 10.1126/science.1177486. Epub 2009 Nov 5. PMID 19892944
- [Background] Ishikawa J, Shimotoyodome Y, Ito S, Miyauchi Y, Fujimura T, Kitahara T, Hase T. Variations in the ceramide profile in different seasons and regions of the body contribute to stratum corneum functions. Arch Dermatol Res. 2013 Mar;305(2):151-62. doi: 10.1007/s00403-012-1286-5. Epub 2012 Sep 18. PMID 22987221